CLINICAL TRIAL: NCT03142724
Title: Assessment of the Biodistribution and Safety of [18F]MNI-968 (Aka PF-06730110) in Healthy Subjects
Brief Title: Assessment of the Biodistribution and Safety of [18F]MNI-968 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-968 Dosimetry
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-968 (Experimental): To assess the safety and tolerability and to determine the radiation dosimetry of [18F]MNI-968.
  Interventions: Drug: [18F]MNI-968

INTERVENTIONS:
Drug: [18F]MNI-968 — Healthy volunteers recruited for the study will undergo a single [18F]MNI-968 injections and PET scans.
  Other Names: PF-06730110

SUMMARY:
The overall goal of this protocol is to evaluate the biodistribution of [18F]MNI-968 as a D1 receptor targeted radiopharmaceutical.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate the biodistribution of [18F]MNI-968 as a D1 receptor targeted radiopharmaceutical. The specific objectives are:

* To determine the radiation dosimetry of [18F]MNI-968
* To assess the safety and tolerability of a single dose of [18F]MNI-968

ELIGIBILITY:
Inclusion Criteria

* The participant is 18 to 55 years old.
* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures

Exclusion Criteria

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject is a currently exposed to nicotine products or had regular nicotine exposure within a six month period, to be verified by urine cotinine screening.
* History of drug or alcohol abuse within 12 months prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during the screening visit.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure does not exceed the effective dose of 50 mSv, equivalent with the acceptable annual limits established by the US Federal Guidelines.
* Pregnancy or women who are breastfeeding, lactating or nursing.
* Unsuitable veins for repeated venipuncture.
* History of immunodeficiency diseases, including a positive HIV test result
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Whole body tomographic PET images will be obtained for 6 healthy volunteers, and reviewed visually for assessment of body organ distribution of radioactivity. | 2 Months
  Volumes of interest (VOI) will be placed on the visually identified source organs, and subsequently used for all the study PET frames. Activity within these volumes of interest is expressed in units of total radioactivity (kBq). Radioactivity will be corrected for body attenuation, but not for decay, and time activity data (TAC) generated for each source organ.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Madonia, PA-C, Principal Investigator — Molecular NeuroImaging, LLC
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://mnimaging.com/